CLINICAL TRIAL: NCT06393387
Title: Retrospective Review of DTG/3TC Versus BIC/F/TAF Across a Multi Clinic Infectious Disease Organization in Southeast United States (REVIVE Study)
Brief Title: Retrospective Review of DTG/3TC Versus BIC/F/TAF Across a Multi Clinic Infectious Disease Organization in Southeast United States
Status: Completed | Type: Observational
Sponsor: Midway Specialty Care Center (Other)
Responsible Party: Principal Investigator, Jennifer Kuretski, Director of Research and Education, Midway Specialty Care Center
Other Study IDs: 222132
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hiv; HIV-1-infection; HIV Infections
Keywords: HIV; Social Determinants of Health; Adherence; Viral Suppression; Percent of Days Covered
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Persons with HIV on DTG/3TC: All data for PWH, initiated on DTG/3TC or BIC/F/TAF, between May 1, 2019 through January 28, 2023, will be collected for purposes of this retrospective study. 400 PWH on DTG/3TC and 400 PWH on BIC/F/TAF, for a total of 800 PWH, will be selected at random for inclusion in this retrospective study.
  Interventions: Drug: DTG/3TC versus BIC/F/TAF
- Persons with HIV on BIC/F/TAF: All data for PWH, initiated on DTG/3TC or BIC/F/TAF, between May 1, 2019 through January 28, 2023, will be collected for purposes of this retrospective study. 400 PWH on DTG/3TC and 400 PWH on BIC/F/TAF, for a total of 800 PWH, will be selected at random for inclusion in this retrospective study.
  Interventions: Drug: DTG/3TC versus BIC/F/TAF

INTERVENTIONS:
Drug: DTG/3TC versus BIC/F/TAF — A new-user, active comparator, retrospective cohort study design will be employed using inverse probability of treatment weighting to adjust for measured confounders. This study will be conducted as a retrospective chart review and the organization's electronic health record (EHR) will be utilized. Subjects identified as having previously been or currently receiving DTG/3TC or BIC/F/TAF will be assessed for eligibility based on inclusion/exclusion criteria. Subject eligibility will be confirmed by the Principal Investigator (PI).

SUMMARY:
This real-world retrospective study describes the clinical efficacy of 2DR (DOVATO® (DTG/3TC)) versus 3DR (BIKTARVY® (BIC/F/TAF)) in PWH, including those with at least 2 social determinants of health indicators, across a multi clinic infectious disease organization in the Southeast United States

DETAILED DESCRIPTION:
3-drug regimens (3DR) have been the foundation of HIV treatment for the last two decades; however, based on more recent data from GEMINI 1 and 2, TANGO, SALSA and STAT clinical trials, 2-drug regimens (2DR), such as dolutegravir/lamivudine, have shown similar efficacy in viral suppression as compared to 3DR1,2,5,6. Furthermore, real-world evidence (RWE) data has reinforced the clinical trial data, showing similar effectiveness outcomes data of DTG/3TC vs. 3DR across ~38,000 people living with HIV, in a variety of sub-populations, including more than 1,200 who are ART naïve. Test and treat strategies have also been successful with both 2DR and 3DR3, but analysis of clinical outcomes, including barriers to resistance as evidenced by viral suppression, in persons with more challenging to treat HIV (PWH), are needed, including PWH with social determinant of health (SDOH) indicators (including but not limited to unstable housing, food insecurity, unemployment, uninsured and/or unstable transportation). PWH may prioritize addressing these needs over adherence to antiretroviral therapy and lower adherence to antiretroviral therapy raises the concern for lack of viral suppression and/or the development of resistance.

A recent study demonstrated that PWH in the United States with 2 or more SDOH indicators were 20% less likely to report excellent adherence in the prior 30 days and 10% less likely to achieve sustained viral suppression in the prior year4 . Furthermore, as HIV disproportionately affects persons of lower socioeconomic status who are experiencing multiple SDOH indicators, identifying ART that can be used to achieve viral suppression in this patient population is essential.

This retrospective study will be performed across a not-for-profit multi-clinic infectious disease organization in the Southeast United States comprising 12 clinics. This multi-clinic infectious disease organization provided care to over 6,000 PWH over the last 5 years. 25% of those PWH identified as cisgender females. 60% of the total PWH were ages 50 years and older. Over 50% of PWH identified their race as a racial and/or ethnic minority.

10 out of 12 clinics are located in 5 of Florida's 6 top counties for prevalence of persons with HIV (Miami-Dade, Broward, Orange, Palm Beach, and Hillsborough Counties). 6 out of 12 clinics provide care for persons with HIV with Ryan White (persons with federal poverty level below 400%). Clinics across the organization provide rapid entry to care for PWH to enter care for the first time (treatment naïve) and/or re-enter care, after being out of care and/or off of ART. The rapid entry to care model also provides the opportunity to review clinical outcomes of PWH starting on either 2DR or 3DR who are re-entering care with an unknown history of resistance.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 18 years and older;
* Diagnosis of HIV-1;
* Have a history of ART consisting of DTG/3TC or BIC/F/TAF, initiated from May 1, 2019 through January 28, 2023;
* Have at least 48 weeks of clinical follow up after initiation of DTG/3TC or BIC/F/TAF; clinical follow-up can include time post-discontinuation of either index regimen;
* Complete data, for HIV-1 RNA viral load at all study time points, including baseline, through 24 weeks and through 48 weeks;
* Received care from a physician, nurse practitioner or physician assistant at the organization

Exclusion Criteria:

* Index regimen is BIC/F/TAF and has a history of ART consisting of DTG+3TC or DTG/3TC;
* Index regimen is DTG/3TC and has a history of ART consisting of BIC/F/TAF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PWH from all 12 sites in Florida across Midway Specialty Care Center.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Viral Suppression | 48 Weeks
  To evaluate the effectiveness of switching treatment to DTG/3TC vs. BIC/F/TAF through 48 weeks in virally suppressed ART experienced individuals with no interruptions in prior therapy.

SECONDARY OUTCOMES:
Viral Suppression | 24 Weeks
  To evaluate the effectiveness of switching treatment to DTG/3TC vs. BIC/F/TAF through 24 weeks in virally suppressed ART experienced individuals with no interruptions in prior therapy.
Viral Suppression | 48 Weeks
  To evaluate the effectiveness of DTG/3TC vs. BIC/F/TAF through 48 weeks in ART naïve individuals (i.e., no prior ART regimen received).
Viral Suppression | 24 Weeks
  To evaluate the effectiveness of DTG/3TC vs. BIC/F/TAF through 24 weeks in ART naïve individuals.
Viral Suppression | 48 Weeks
  To evaluate the effectiveness of DTG/3TC vs. BIC/F/TAF through 48 weeks in ART experienced individuals who are returning to care (i.e., previous ART therapy received but not in the last month).
Viral Suppression | 24 Weeks
  To evaluate the effectiveness of DTG/3TC vs. BIC/F/TAF through 24 weeks in ART experienced individuals who are returning to care.
Clinical Characteristics of Persons with HIV | Baseline
  To describe the baseline demographics and clinical characteristics of individuals on DTG/3TC and BIC/F/TAF by the following sub-groups: (1) Virally suppressed, (2) ART experienced individuals, & (3) ART naïve individuals ART experienced individuals who are returning to care
Tolerability | 24, 48 Weeks
  To assess the tolerability (i.e., all drug-related adverse reactions (ARs) as per label) of DTG/3TC vs. BIC/F/TAF through 24 weeks and 48 weeks by the following sub-groups: (1) Virally suppressed ART experienced individuals, (2) ART naïve individuals & (3) ART experienced individuals who are returning to care.
Treatment Discontinuation | 24, 48 Weeks
  To assess treatment discontinuations (i.e., withdrawals due to drug-related ARs) of DTG/3TC vs. BIC/F/TAF through 24 weeks and 48 weeks by the following sub-groups: (1) Virally suppressed ART experienced individuals, (2) ART naïve individuals, (3) ART experienced individuals who are returning to care.

OTHER OUTCOMES:
Viral Suppression | 48 Weeks
  To evaluate the effectiveness of switch to DTG/3TC vs. BIC/F/TAF through 48 weeks in virally suppressed ART experienced individuals by the following sub-groups: (1) At least 2 social determinants of health, (2) Cisgender females, (3) Aged 50 years or older, & (4) Unknown baseline resistance (defined as absence of genotypic documentation on resistance at point of index treatment initiation)
Viral Suppression | 48 Weeks
  To evaluate the effectiveness of DTG/3TC vs. BIC/F/TAF through 48 weeks in ART naïve individuals by the following sub-groups: (1) At least 2 social determinants of health, (2) Baseline VL > 100,000 copies/mL, (3) Baseline VL > 400,000 copies/mL, (4) Baseline absolute CD4 count of <200 cells/m3, (5) Cisgender females, (6) Aged 50 years or older, & (7) Unknown baseline resistance
Viral Suppression | 48 Weeks
  To evaluate the effectiveness of DTG/3TC vs. BIC/F/TAF through 48 weeks in ART experienced individuals who are returning to care (i.e., previous ART therapy received but not in the last month) by the following sub-groups: (1) At least 2 social determinants of health, (2) Baseline VL > 100,000 copies/mL, (3) Baseline VL > 400,000 copies/mL, (4) Baseline absolute CD4 count of <200 cells/m3, (5) Cisgender females, (6) Aged 50 years or older, & (7) Unknown baseline resistance
Weight Change | 48 Weeks
  To describe and compare the change in weight / BMI of DTG/3TC vs. BIC/F/TAF through 48 weeks by the following sub-groups: (1) Virally suppressed ART experienced individuals, (2) ART naïve individuals, & (3) ART experienced individuals who are returning to care
Change in Absolute CD4 and CD4/CD8 Ratio | 48 Weeks
  To describe and compare immune recovery from baseline indicated by change in CD4 cell count and CD4/CD8 ratios of DTG/3TC vs. BIC/F/TAF through 48 weeks by the following sub-groups: (1) Virally suppressed ART experienced individuals, (2) ART naïve individuals, & (3) ART experienced individuals who are returning to care
Viral Suppression | 24, 48 Weeks
  To evaluate the effectiveness of DTG/3TC vs. BIC/F/TAF as defined by the proportion of ART experienced individuals who are returning to care with HIV-1 RNA level <20 copies/mL through 24 weeks and 48 weeks
Persistence on DTG/3TC versus BIC/F/TAF | 24, 48 Weeks
  To describe available self-reported persistence to DTG/3TC vs. BIC/F/TAF regimens through 24 weeks and 48 weeks, by the following subgroups: (1) Virally suppressed ART experienced individuals, (2) ART naïve individuals, & (3) ART experienced individuals who are returning to care

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kuretski, DNP, Principal Investigator — Midway Specialty Care Center
Locations (1):
- Midway Specialty Care Center, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cahn P, Madero JS, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man C, Currie A, Underwood M, Tenorio AR, Pappa K, Wynne B, Fettiplace A, Gartland M, Aboud M, Smith K; GEMINI Study Team. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferiority, phase 3 trials. Lancet. 2019 Jan 12;393(10167):143-155. doi: 10.1016/S0140-6736(18)32462-0. Epub 2018 Nov 9. PMID 30420123
- [Background] Cahn P, Sierra Madero J, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man CY, Urbaityte R, Brandon DJ, Underwood M, Pappa KA, Curtis L, Smith KY, Gartland M, Aboud M, van Wyk J, Wynne B. Three-year durable efficacy of dolutegravir plus lamivudine in antiretroviral therapy - naive adults with HIV-1 infection. AIDS. 2022 Jan 1;36(1):39-48. doi: 10.1097/QAD.0000000000003070. PMID 34534138
- [Background] Menza TW, Hixson LK, Lipira L, Drach L. Social Determinants of Health and Care Outcomes Among People With HIV in the United States. Open Forum Infect Dis. 2021 Jun 22;8(7):ofab330. doi: 10.1093/ofid/ofab330. eCollection 2021 Jul. PMID 34307729
- [Background] van Wyk J, Ajana F, Bisshop F, De Wit S, Osiyemi O, Portilla Sogorb J, Routy JP, Wyen C, Ait-Khaled M, Nascimento MC, Pappa KA, Wang R, Wright J, Tenorio AR, Wynne B, Aboud M, Gartland MJ, Smith KY. Efficacy and Safety of Switching to Dolutegravir/Lamivudine Fixed-Dose 2-Drug Regimen vs Continuing a Tenofovir Alafenamide-Based 3- or 4-Drug Regimen for Maintenance of Virologic Suppression in Adults Living With Human Immunodeficiency Virus Type 1: Phase 3, Randomized, Noninferiority TANGO Study. Clin Infect Dis. 2020 Nov 5;71(8):1920-1929. doi: 10.1093/cid/ciz1243. PMID 31905383
- [Background] Maggiolo F, Valenti D, Teocchi R, Comi L, Filippo ED, Rizzi M. Adherence to and Forgiveness of 3TC/DTG in a Real-World Cohort. J Int Assoc Provid AIDS Care. 2022 Jan-Dec;21:23259582221101815. doi: 10.1177/23259582221101815. PMID 35695220
- [Background] Maggiolo F , MD, Valenti D , BSc, Teocchi R , BSc, Comi L , MD, Di Filippo E , MD, Rizzi M , MD. Real World Data on Forgiveness to Uncomplete Adherence to Bictegravir/ Emtricitabine/Tenofovir Alafenamide. J Int Assoc Provid AIDS Care. 2022 Jan-Dec;21:23259582221140208. doi: 10.1177/23259582221140208. PMID 36423244
- [Background] Rolle CP, Berhe M, Singh T, Ortiz R, Wurapa A, Ramgopal M, Leone PA, Matthews JE, Dalessandro M, Underwood MR, Angelis K, Wynne BR, Merrill D, Nguyen C, van Wyk J, Zolopa AR. Dolutegravir/lamivudine as a first-line regimen in a test-and-treat setting for newly diagnosed people living with HIV. AIDS. 2021 Oct 1;35(12):1957-1965. doi: 10.1097/QAD.0000000000002979. PMID 34115650
- See also: Related Info — https://medinfo.gsk.com/5f95dbd7-245e-4e65-9f36-1a99e28e5bba/ea58ece8-e706-4777-b8f8-eebe4eaa4b79/ea58ece8-e706-4777-b8f8-eebe4eaa4b79_viewable_rendition__v.pdf?medcommid=REF--ALL-004495